CLINICAL TRIAL: NCT06830733
Title: Phase II, Multicenter, Open-label, Prospective, Non-randomized Study to Evaluate the Safety and Efficacy of ARI0002h, a CAR-T Cell Against BCMA, for the Initial Treatment of Patients With Primary Plasma Cell Leukaemia
Brief Title: Study to Evaluate the Safety and Efficacy of ARI0002h, for the Initial Treatment of Patients With Primary Plasma Cell Leukaemia
Acronym: GEM-PLASMACAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-515053-21-00
Record Dates: First submitted 2024-11-20; First posted 2025-02-17 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-02

CONDITIONS: Leukemia, Plasma Cell
MeSH Terms: conditions — Leukemia, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARI0002h (Experimental): ARI0002 will be administered intravenously in two doses. First dose will b e a fractionated infusion of three doses of the investigational medicinal product (day 0: 10% dose, day 3: 30% dose, day 7: 60% dose), and a second adminsitration as a single dose at 2 months after the first in those patients who have achieved at least a minimal response, have not presented PCL progression after the first infusion or serious complications after the first infusion.
  Interventions: Genetic: ARI0002h

INTERVENTIONS:
Genetic: ARI0002h — * Treatment with ARI0002h cells
  * Other names: CARTBCMA_J22.9-h:CD8TM:4-1BB:CD3. Adult differentiated autologous T cells from peripheral blood, expanded and transduced with a lentivirus to express a chimeric antigen receptor with anti-BCMA (TNFRSF17) specificity conjugated to the 4-1BB co-stimulatory domain and the CD3z signalling domain that has been humanized.

SUMMARY:
Phase II, pilot, open-label, prospective, multicenter, non-randomized study to evaluate the safety and efficacy of ARI0002h (cesnicabtagene autoleucel) in 20 patients with newly diagnosed primary plasma cell leukemia (PCL).

The study population is patients between 18 and 75 years of age with newly diagnosed primary plasma cell leukemia (pPCL), with a life expectancy of more than 3 months.

The primary objective is to assess the safety and efficacy of CARTBCMA ARI0002h (cesnicabtagene autoleucel) after initial treatment to induce response in patients with newly diagnosed primary plasma cell leukaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 75 years old diagnosed with newly diagnosed primary plasma cell leukemia (the presence of 5% or more circulating plasma cells in peripheral blood smears in patients otherwise diagnosed with symptomatic multiple myeloma), according to International Myeloma Working Group (IMWG).
2. Disease measurable at diagnosis by monoclonal component in serum or urine, or by free light chains in serum according to the eligibility criteria for clinical trials of the "International Myeloma Working Group".
3. ECOG Performance Status from 0 to 2
4. Life expectancy greater than 3 months.
5. Adequate venous access and absence of contraindications for lymphoapheresis.
6. Patients who, after being informed, give their consent by signing the Informed Consent Document.
7. Up to two cycles of previous treatment for symptomatic control will be allowed before inclusion.

Exclusion Criteria:

1. No previous treatments, except for induction therapy for primary plasma cell leukemia.
2. Administration of any anti-BCMA therapy as part of induction
3. Not having achieved at least a minimal response with induction treatment (IMWG criteria)
4. Absolute lymphocyte count <0.1x109/L
5. Active immunosuppressive therapy except for prednisone 10 mg/day (or equivalent).
6. Any other concomitant neoplasia, unless it has been in complete remission for 3 years or longer, except for non-melanoma skin cancer or completely resected in situ carcinoma.
7. Active infection requiring treatment.
8. Active HIV, HBV, or HCV infection.
9. Uncontrolled medical illness
10. Severe organ impairment that meets any of the following criteria: EF<40%, DLCO <40%, GFR <30 ml/min, bilirubin >3 times the upper limit of normality (unless due to Gilbert syndrome)
11. Previous diagnosis of symptomatic AL amyloidosis,
12. Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at the screening phase.
13. Women of childbearing potential, including those whose last menstrual cycle was in the year prior to screening, who are unable or unwilling to use highly effective contraceptive methods* from the beginning of the study to completion of the study.
14. Men who are unable or unwilling to use highly effective contraceptive methods* from the beginning of the study to completion of the study.
15. Contraindication to receive lymphodepletive chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 months after the first infusion
  Overall response rate (ORR) during the initial 3 months after the first infusion (at least presenting a partial response according to the International Myeloma Working Group criteria).
Rate of patients who develop cytokine release syndrome and/or neurological toxicity | 30 days after CARTBCMA administration
  Rate of patients who develop cytokine release syndrome and/or neurological toxicity in the first 30 days after CARTBCMA administration, according to the criteria and grading defined in the international consensus document

SECONDARY OUTCOMES:
Duration of response | From day 28 after infusion to study completion, an average of 24 months
  Duration of response calculated from the time of first disease evaluation
Response rates | During the first year after administration
  Response rates
Complete response rate | at 3, 6, and 12 months after the first infusion
  Complete response rate
Overall response rate | at 6, and 12 months after the first infusion
  Overall response rate
Time to complete response | through study completion, an average of 24 months
  Time to complete response
Time to best response | through study completion, an average of 24 months
  Time to best response
MRD negative rate in bone marrow | at 3, 6 12 and 24 months
  MRD negative rate in bone marrow by flow cytometry
Response rate of extramedullary disease | at 3, 6 and 12 months.
  Response rate of extramedullary disease by PET-CT
Progression-free survival | through study completion, an average of 24 months
  defined as the time between administration of ARI0002h and disease progression or death. Patients who are alive and in complete remission will be censored at the time of the last follow-up.
Progression-free survival at 12 months after the first administration | 12 months
  Progression-free survival at 12 months after the first administration, defined as the time elapsed between the administration of ARI0002h and disease progression or death. Patients who are alive and in complete remission will be censored at the time of the last follow-up.
Overall survival | through study completion, an average of 24 months
  Overall survival, defined as the time between infusion of ARI0002h and death of the patient from any cause. Living patients will be censored at the time of last follow-up.
Presence of infusion reactions | through study completion, an average of 24 months
  Presence of infusion reactions, understood as the appearance of any of the following symptoms after the intravenous administration of CARTBCMA: cardiac events, chills, dyspnea, fatigue, sudden hypertension, hypotension, nausea, pain, fever, rash or urticaria.
Tumour lysis syndrome | through study completion, an average of 24 months
  Tumour lysis syndrome
Cytokine release syndrome | through study completion, an average of 24 months
  Cytokine release syndrome. According to the criteria and grading defined in the international consensus document
Neurological toxicity | through study completion, an average of 24 months
  Neurological toxicity according to the criteria and grading defined in the international consensus document (Lee, Santomasso et al. 2019)
Presence of prolonged cytopenias | between 4 weeks after infusion and study completion
  Presence of prolonged cytopenias, defined as a grade 4 decrease in peripheral blood neutrophil or platelet counts for more than 4 weeks after infusion.
Quality of life of patients | during the first year after infusion
  Quality of life during the first year after infusion according to the Quality of life questionnaire 2008 EuroQol Group EQ-5D

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Clínica Universitaria de Navarra, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Asistencial Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Clinic Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No